CLINICAL TRIAL: NCT07011602
Title: INTEGRATED CHILDHOOD ACTIVITY AND NUTRITION (ICAN) STUDY
Acronym: ICAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: United States Department of Agriculture - National Institute of Food and Agriculture (USDA-NIFA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0625
Record Dates: First submitted 2025-06-05; First posted 2025-06-09 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-06

CONDITIONS: Achievement; Weight Change; Cognition; Fitness; Nutrition Status
Keywords: brain, exercise, carotenoids, body composition
MeSH Terms: conditions — Body Weight Changes; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): 8-week Physical Activity and Nutrition
  Interventions: Behavioral: 8-week Physical Activity and Nutrition Program
- Control (No Intervention): Waitlist Control

INTERVENTIONS:
Behavioral: 8-week Physical Activity and Nutrition Program — Participants will be enrolled in an 8-week (Monday-Friday) daily physical activity program where treatment group participants will receive daily physical activity via organized games and daily lutein (6mg/d) snacks.
  Arms: Treatment Group

SUMMARY:
This study is a multi-functional integrated research and education project to prevent losses in academic achievement, cognitive function, and behavioral health among at-risk youth. The study tests the effects of a 8-week nutrition and physical activity-based program (Integrated Childhood Activity and Nutrition [ICAN]) to prevent summer learning loss. Outcomes include standardized academic achievement as well as executive function among 6-10-year-olds affected by poverty. The nutrition component of the intervention involves daily consumption of a snack containing the carotenoid lutein, typically found in high quantities in green leafy vegetables. The physical activity components will involve group games or activities.

DETAILED DESCRIPTION:
During the summer period it is estimated that children, especially those from impoverished settings, could lose up to 30% of learning gained during the school year. Additionally, the loss in learning accompanied by increased risk for obesity. Children's dietary intake, particularly of nutrient-dense dark green leafy vegetables, has persistently fallen below dietary recommendations. Similarly, there has been a decline in children's aerobic fitness since the 1970s. Despite consistent and widespread efforts, there has been limited progress in improving children's dietary habits, habitual physical activity engagement, and reducing child obesity. One reason for this perpetual challenge is that educational and intervention efforts typically occur during the school year. However, it is the summer, not the school year, when accelerated increases in body fat and decline in diet quality and physical activity tend to occur. Student summer learning loss, a phenomenon commonly referred to as the summer slide, is the loss of academic knowledge and/or skills during the summer. Students' achievement scores decline over the summer by one month's worth of school-year learning instruction. Additionally, these effects are more pronounced black and Latino students who not only tend to gain less over the school year but exhibit greater learning loss in the summer, compared to white students. This is at least in part because during summer, fewer opportunities exist for children from low-income households to access healthy structured programs. Therefore, efficacious nutrition and physical activity-based programs are critically needed, especially during summer, a period of vulnerability among children affected by poverty.

This work will conduct an 8-week physical activity and nutrition randomized controlled trial among children during the summer period. The specific aims are outlined below.

Specific Aim 1: To investigate the effects of combining an 8-week lutein intervention (6mg lutein/day) with a social emotional learning (SEL)-framed physical activity summer intervention (ICAN) on improving academic achievement and cognition among school children (6-11-year-olds) affected by poverty.

Specific Aim 2: To investigate the effects of the ICAN program on improvement in carotenoid status and implications for academics and cognition in 6-11-year-olds from impoverished settings.

Specific Aim 3: To investigate ICAN intervention effects on weight status and adiposity.

ELIGIBILITY:
Inclusion Criteria:

* Parental/guardian consent
* Child assent
* Child participant is between the chronological age of 6-11 years.
* Child participant is considered economically or educationally disadvantaged (e.g., eligible for Supplemental Nutritional Assistance Program [SNAP] and/or qualifies for free-and-reduced lunch.
* Child participant must have 20/20 or corrected 20/20 vision.
* Child participant absent of cognitive or neurological disorder (e.g., autism spectrum disorder)

Exclusion Criteria:

* Parental/guardian does not provide consent
* Child non-assent
* Child participant chronological age when enrolling into the iCANS program falls below 6 or above 11 years of age
* Child participant is not eligible for SNAP or does not qualify for free-and-reduced lunch.
* Child participant does not have 20/20 or corrected 20/20 vision.
* Presence of cognitive or neurological disorder (e.g., autism spectrum disorder)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Academic Achievement | Baseline vs. 8 week Post-test
  Composite score on the standardized Kaufman Test of Academic and Educational Achievement 3-(KTEA-3)

SECONDARY OUTCOMES:
Attentional Inhibition | Baseline vs. 8-week Post-test
  Flanker Task Accuracy (%)
Attentional Inhibition | Baseline vs. 8-week Post-test
  Flanker Reaction Time (ms)
Attentional Resource Allocation | Baseline vs. 8 week Post-test
  P3 Event-related potential amplitude (mv)
Processing Speed | Baseline vs. 8 week Post-test
  P3 Event-related potential latency (ms)
Retinal Xanthophylls | Baseline vs. 8 week Post-test
  Macular Pigment Optical Density
Skin Carotenoids | Baseline vs. 8 week Post-test
  Veggiemeter Score
Weight status | Baseline vs. 8 week Post-test
  BMI-for-age Percentile
Adiposity | Baseline vs. 8 week Post-test
  %Fat assessed by bioelectric impedance
Nutrition Literacy | Baseline vs. 8 week Post-test
  Nutrition Literacy Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Bloomington Public Schools District 87, Bloomington, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided